CLINICAL TRIAL: NCT06418282
Title: An Open-label, Multi-center, Prospective VA Study to Evaluate the Effectiveness and Health Economics of a Novel Portable Non-Pneumatic Active Compression Device (NPCD) for Lymphedema/Phlebolymphedema
Brief Title: Clinical Study to Evaluate the Effectiveness and Health Economics of a Novel Portable Non-Pneumatic Active Compression Device (NPCD) for Lymphedema/Phlebolymphedema
Acronym: GRANDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koya Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCT 013 (GRANDE)
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Phlebolymphedema; Lymphedema; Chronic Venous Insufficiency
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dayspring, Non-Pneumatic Active Compression Device (NPCD) (Experimental): The Dayspring, an Non-Pneumatic Active Compression Device (NPCD) Active Wearable Compression Device is an FDA cleared calibrated active gradient pressure compression garment that is segmental and programmable and applies controlled sequential pressure from the distal to proximal-end of the limb in a cyclic manner.
  Interventions: Device: Dayspring

INTERVENTIONS:
Device: Dayspring — NPCD

SUMMARY:
An open-label, multi-center, prospective VA study to evaluate the effectiveness and health economics of a Novel Portable Non-Pneumatic Active Compression Device (NPCD) for lymphedema/phlebolymphedema

DETAILED DESCRIPTION:
An open-label, multi-center, prospective VA study to evaluate the effectiveness and health economics of a Novel Portable Non-Pneumatic Active Compression Device (NPCD) for lymphedema/phlebolymphedema

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Capable and willing to sign the informed consent and deemed capable of following the study protocol
* Subjects must have a diagnosis of unilateral or bilateral lower extremity edema or lower extremity lymphedema/phlebolymphedema as a consequence of chronic venous insufficiency
* Subjects who have medical clearance using diagnostic confirmation through venous duplex to rule out DVT and superficial/deep reflux

Exclusion Criteria:

* Inability or unwillingness to participate in all aspects of study protocol and/or inability to provide informed consent
* Individuals with a history or presence of a systemic disorder or condition that could place the subject at increased risk from sequential compression therapy
* Subjects must not have any diagnosed cognitive or physical impairment that would interfere with the use of the device
* Non-ambulatory individuals
* Female: BMI > 34 (5'4", 200 lbs.)
* Male: BMI > 34 (5'9", 230 lbs.)
* (Max circumference at patella 58 cm; Max circumference at gluteal fold 75 cm)
* Diagnosis of lipedema
* Diagnosis of active or recurrent cancer (< 3 months since completion of chemotherapy, radiation therapy or primary surgery for the cancer)
* Diagnosis of acute infection (in the last four weeks)
* Diagnosis of active/open wound/ulcer
* Diagnosis of acute thrombophlebitis (in last 2 months)
* Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 6 months
* Diagnosis of pulmonary edema
* Diagnosis of congestive heart failure (uncontrolled/uncompensated)
* Diagnosis of chronic kidney disease with acute renal failure
* Diagnosis of epilepsy
* Subjects with poorly controlled asthma
* Any condition where increased venous and lymphatic return is undesirable
* Women who are pregnant, planning a pregnancy or nursing at study entry
* Participation in any clinical trial of an investigational substance or device during the past 30 days

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Lymphedema Overall Quality of Life and Patient Survey | 6 months
  The Lymphedema Quality of Life Questionnaire (LYMQOL), a validated disease-specific QoL tool, is also administered at baseline and month 3. Overall QoL is scored on a single item by the patient on a scale of 1-10. The outcome measure is assessed as a difference or change from baseline LYMQOL at day zero and month 6
Cost comparison between NPCD and historical reference (as reflected by hospital/resource utilization related to adverse events) | 6 months
  Cost comparison between NPCD and historical reference (as reflected by hospital/resource utilization related to adverse events)
Mobility (daily steps using a pedometer) | 6 months
  Mobility (daily steps using a pedometer)

SECONDARY OUTCOMES:
Lower extremity edema response (limb girth reduction) | 6 months
  Lower extremity edema response (limb girth reduction)
LE Functional Index (LEFI) | 6 months
  LE Functional Index (LEFI)
Venous Clinical Severity Score (VCSS) | 6 months
  Venous Clinical Severity Score (VCSS) scored on severity from None (0), Mild (1), Moderate (2) to Severe (3). Higher score means a worse outcome
Safety/Adverse Events | 6 months
  As assessed by reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Glenn Jacobowitz, New York, New York, United States